CLINICAL TRIAL: NCT01444508
Title: Effect of Colloid Versus Crystalloid on Coagulation in Elective Urological Surgery
Brief Title: Effect of Colloid Versus Crystalloid on Coagulation
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: K. C. Rasmussen (Other)
Responsible Party: Sponsor-Investigator, K. C. Rasmussen, MD, specialist in surgery and research fellow, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2011-003270-80
Record Dates: First submitted 2011-09-10; First posted 2011-09-30 (Estimated); Last update posted 2013-12-13 (Estimated); Status verified 2013-12

CONDITIONS: Bloodloss
MeSH Terms: interventions — HES 130-0.4

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- crystalloid (Active Comparator)
  Interventions: Drug: Ringer-lactate "SAD"
- colloid (Placebo Comparator)
  Interventions: Drug: HES 130/04

INTERVENTIONS:
Drug: Ringer-lactate "SAD" — Lactated Ringer's is administrated intravenously in the dosis of max. 35 ml/kg during the operation after securing normovolaemia with Nexfin Monitor at induction of the anaesthesia: if bolus infusion of 200 ml increases stroke volume more than 10 % the patient is not assumed normovolaemic and bolus infusions are repeated until normovolaemic status is achieved.
  Other Names: Ringer-laktat "SAD", B 05 BB 01, Amgros A/S.
  Arms: crystalloid
Drug: HES 130/04 — Voluven is administered intravenously in the doses of max. 35 ml/kg during the operation. Normovolaemia is achieved in the same way as described in intervention by Ringer-lactate "SAD".
  Other Names: Voluven, HES 130/04, B 05 AA 07, Fresenius Kabi A/S.
  Arms: colloid

SUMMARY:
In order to reduce bloodloss and need for transfusion to investigate the effect of colloid and crystalloid on coagulation assuming no difference between the groups.

ELIGIBILITY:
Inclusion Criteria:

* Patient more than 18 years old
* Indication for elective post-renal operation including cystectomy
* Patient without anticoagulative, acetylsalicylic acid or NSAID treatment for the last 5 days.

Exclusion Criteria:

* Intracerebral bleeding, manifest cardiac insufficient, renal insufficient demanding dialysis, hepatic or coagulation diseases
* Pregnant or nursing
* Allergic
* Disturbance in electrolytes
* Patient under committee
* Patient joining another trial interfering the actual trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2011-09; Primary Completion 2013-04 (Actual); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Effect of colloid versus crystalloid on laboratory coagulation. | 5-7 hours
  Coagulation is analysed in bloodsamples before, during (10 minutes post cystectomia), at the end of the operation and 2 hours later on.
  The bloodsamples are analysed by thromboelastography (5000 series TEG analyzer, Haemoscope Corporation, Niles IL, USA) besides the classic coagulation parametres: platelet count, INR, Fibrinogen, APTT, D-dimer and Haemoglobin, Amylase and Creatinin.

SECONDARY OUTCOMES:
Effect of colloid versus crystalloid on the amount of bloodloss | 5-7 hours
  The water balance inclusive the amount of bloodloss is registrated at the end of the operation and 2 hours later on.

CONTACTS AND LOCATIONS:
Locations (1):
- Rigshospitalet, Copenhagen, Denmark

REFERENCES:
- [Derived] Rasmussen KC, Johansson PI, Hojskov M, Kridina I, Kistorp T, Thind P, Nielsen HB, Ruhnau B, Pedersen T, Secher NH. Hydroxyethyl starch reduces coagulation competence and increases blood loss during major surgery: results from a randomized controlled trial. Ann Surg. 2014 Feb;259(2):249-54. doi: 10.1097/SLA.0000000000000267. PMID 24100337